CLINICAL TRIAL: NCT02163278
Title: A Double-blind, Randomized, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DBPR108 in Healthy Male Subjects
Brief Title: A Multiple Ascending Dose Phase I Study of DBPR108 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: DBPR108-102
Record Dates: First submitted 2014-06-06; First posted 2014-06-13 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: DBPR108; DPP4; Diabetes; Glucagon-like peptide-1 (GLP-1); Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — DBPR108

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DBPR108 (Experimental)
  Interventions: Drug: DBPR108
- matching placebo (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: DBPR108 — DBPR108 capsules in four doses beginning at 25 mg and rising to 600 mg.
  Arms: DBPR108
Drug: matching placebo — Matching placebo capsules in four doses beginning at 25 mg and rising to 600 mg.
  Arms: matching placebo

SUMMARY:
The study is being performed to assess the safety, tolerability, and pharmacokinetic (PK) and pharmacodynamic (PD) properties of multiple oral doses of DBPR108 in healthy male subjects.

DETAILED DESCRIPTION:
This study represents the administration of dipeptidyl peptidase 4 (DPP4) inhibitor DBPR108 to humans to evaluate the safety, tolerability, and pharmacokinetic (PK) and pharmacodynamic (PD) properties following multiple oral doses in healthy subjects.

DPP4 is a validated drug target for the treatment of human type 2 diabetes. Objectives of the study will be to assess the safety and tolerability, PKs and PDs of DBPR108 at steady state after administration of multiple oral doses to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male with suitable veins for cannulation or repeated venipuncture, and must be able to swallow the investigational product intact.
* Aged between 20 and 45 years (inclusive) at the screening visit.
* Able to provide written informed consent and willing to comply with the study protocol procedures and restrictions.

Exclusion Criteria:

* Has a body weight less than 50 kg and/or body mass index (BMI) less than 18.5 kg/m2 or greater than or equal to 24 kg/m2 at the screening visit. Body mass index is determined as total body weight/height2 (kg/m2).
* Has a creatinine clearance (Ccr) less than 80 mL/min at screening.
* Is not in good general health as judged by the Investigator based on routine medical history, vital signs, physical examination, ECG, laboratory tests, and urinalysis at the screening visit or at admission on Day -1. Normal ECG includes (1) sinus rhythm, (2) pulse rate between 45 and 90 bpm, (3) Corrected QT (QTc) interval equal to or less than 450 ms (corrected cf Bazett 1920), (4) QRS interval less than 110 ms, (5) PR interval less than 200 ms, and (6) morphology consistent with healthy cardiac conduction and function.
* Is not normoglycemic defined as fasting glucose at less than 70 mg/dL (3.9 mmol/L) and greater than 99 mg/dL (5.5 mmol/L), based on the laboratory tests at screening or at admission on Day -1, or has known diabetes or impaired glucose tolerance (Re-testing of fasting glucose on the same sample collected from the subject with initial fasting glucose value of 100-105 mg/dL on Day -1 is acceptable. However, if the re-testing fasting glucose value is still greater than 99 mg/dL, the subject shall be excluded and considered as screen-failure).
* Has a platelet count less than 150,000/μL.
* Uses any antihyperglycemic agents at screening or at admission on Day -1.
* Has a history or presence of any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs at the screening visit or at admission on Day -1.
* Has a clinically significant psychiatric, renal, hepatic, cardiovascular, gastrointestinal, or neurologic disease at screening or at admission on Day -1.
* Is a smoker and/or has used nicotine-containing products within the last 6 months prior to the screening for the current study and/or has a history of alcohol abuse.
* Has donated blood or participated in another clinical study within 8 weeks before Day -1.
* Excessive intake of caffeine-containing drinks or food (i.e., coffee, tea, chocolate, PAOLYTA B Liq, WHISBIH Liq, or cola [more than 6 units of caffeine per day]). One caffeine unit is contained in the following items: 1 (177.4 mL) cup of coffee, 2 (354.9 mL) cans of cola, 1 (354.9 mL) cup of tea, ½ (118.3 mL) cup of energy drink (e.g., PAOLYTA B Liq or WHISBIH Liq), or 3 oz of chocolate.
* Use of drugs with cytochrome P450 enzyme-inducing or
* inhibiting properties within 4 weeks prior to the first administration of investigational product.
* Has used prescription or nonprescription medication (except for occasional use of paracetamol or nasal spray) or herbal remedies or vitamins or minerals within 2 weeks or 5 half-lives of the drug, whichever is longer, prior to dosing until end of study.
* Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of investigational product.
* Male subjects who are unwilling to use barrier contraception in addition to having their partner use another method of contraception, for the duration of the study and for 3 months after dosing.
* Has a positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV).
* Has received a blood transfusion and/or has HCV infection.
* Positive result on screening for drugs of abuse, alcohol, or cotinine (nicotine) at screening or on Day -1.
* Involved in the planning or conduct of the study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Each subject will be followed for the duration of 6 hospital stays, an expected average of 5 weeks

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 33 time points during 12 days (including measurements before dosing)
  PK parameters are including: Cmax, Cmin, Cavg, Cmin,i , Tmax, Tlast, t1/2, AUCτ, AUC0-t, AUC0-inf, % Fluctuation, Apparent body clearance following extravascular dosing (CL/F), Vz/F, Aet1-t2, Ae0-t, fe0-t, Renal clearance (CLR), Accumulation index (AI) and Accumulation ration (AR)
Pharmacodynamic parameters | 34 time points during 10 days (including measurements before dosing)
  PD parameters are including: Emax, Emin, Time to maximum effect (TEmax), TEmin, Area under the response versus time curve during a dosing interval ( AUECτ) and Area under the response versus time curve from time zero to the time of last quantifiable response (AUEC0-t)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University - Taipei Medical University Hospital, Taipei, Taiwan